CLINICAL TRIAL: NCT00295295
Title: Mechanical Intervention in Children With Cerebral Palsy
Brief Title: Vibration Intervention to Improve Bone and Muscle in Children With Cerebral Palsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Tishya Wren, Principal Investigator, Children's Hospital Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1R21AR051564 (NIH); R21AR051564 (NIH); 1R21AR051564 (NIH)
Record Dates: First submitted 2006-02-21; First posted 2006-02-23 (Estimated); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Cerebral Palsy
Keywords: vibration; bone density
MeSH Terms: conditions — Cerebral Palsy | interventions — Standing Position

ARMS (2):
- Vibration (Experimental): High frequency, low magnitude vibration at 30 Hz, 10 min/day using vibrating platform from Juvent Medical Inc.
  Interventions: Device: High frequency, low magnitude vibration
- Standing (Active Comparator): Standing 10 min/day
  Interventions: Other: Standing

INTERVENTIONS:
Device: High frequency, low magnitude vibration — High frequency, low magnitude vibration at 30 Hz, 10 min/day using vibrating platform from Juvent Medical Inc.
  Arms: Vibration
Other: Standing — Standing 10 min/day
  Arms: Standing

SUMMARY:
Cerebral palsy is a group of disorders characterized by lack of coordination in the muscles, loss of movement, and speech disturbances. These disorders are caused by injuries to the brain that occur during fetal development or near the time of birth. The purpose of this study is to determine the effects of high frequency, low magnitude vibration on bone and muscle in children with cerebral palsy.

DETAILED DESCRIPTION:
The extent of bone mass built up during childhood and adolescence is the most important determinant of osteoporosis later in life. Some disabled children, such as those with cerebral palsy, are particularly vulnerable to low bone mass accumulation due to decreased mobility and weight-bearing. These children also have poor muscle strength and control, which limits function and contributes to the lack of mechanical stimulation needed to build bone mass. The most common treatment for these children is physical therapy, which is time- and labor-intensive and may not be adequately available to them. Whole body vibration has shown promise as an alternative method for stimulating increases in bone mass and improvements in muscle. The purpose of this study is to evaluate the effects of high frequency, low magnitude vibration on bone and muscle in children with cerebral palsy. This intervention may be useful as a noninvasive, nonpharmacological treatment for low bone mass and poor muscle function in these children.

This study will last 1 year. All participants will visit the hospital 3 times, at study entry and Months 6 and 12. At each visit, height and weight will be measured, muscle strength and balance will be tested, and bones and muscles in the spine and lower leg will be imaged with computed tomography (CT), a special x-ray machine. Participants will be randomly assigned to one of two groups. For this study, all participants will be asked to stand for 10 minutes every day for 1 year. For Group 1, a vibrating platform will be used for the 10-minute standing sessions during the first half of the study but not during the second half of the study. For Group 2, this will be reversed and the vibrating platform will not be used during the first half of the study but will be used during the second half of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral palsy
* Low vertebral bone density
* Able to stand for 10 minutes with handheld support
* Parent or guardian willing to provide informed consent

Exclusion Criteria:

* Surgery, casting, or receipt of botulinum toxin in the 12 months prior to study entry
* Planned surgery, casting, or receipt of botulinum toxin in the 12 months after study entry
* Metal rods or plates in tibia or lumbar spine
* Severe scoliosis (greater than 20 degrees) or bowing of tibia
* Medical condition other than cerebral palsy affecting bone or muscle
* Require corticosteroids or seizure medication (phenytoin)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34
Dates: Start 2004-09; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Vertebral bone density | Measured at Month 12
Tibia bone density | Measured at Month 12
Tibia cross-sectional area | Measured at Month 12

SECONDARY OUTCOMES:
Calf muscle strength | Measured at Month 12
Balance test | Measured at Month 12
  Clinical balance test used by California Children's Services, Los Angeles County Medical Therapy Units

CONTACTS AND LOCATIONS:
Overall Officials: Tishya A.L. Wren, PhD, Principal Investigator — Children's Orthopaedic Center, Children's Hospital Los Angeles, and Departments of Orthopaedics and Radiology, Keck School of Medicine, Department of Biomedical Engineering, School of Engineering, University of Southern California
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States